CLINICAL TRIAL: NCT03326739
Title: Ultrasound Guided Versus Landmark Guided Arterial Line Placement by Emergency Medicine Interns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 24642
Record Dates: First submitted 2017-10-17; First posted 2017-10-31 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Vascular Access Complication

STUDY DESIGN:
Who Masked: Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound Guided A-Line Placement (Active Comparator): Patients in this group will have ultrasound guided arterial line placement.
  Interventions: Procedure: Arterial Line Placement
- Landmark Guided A-line Placement (Active Comparator): Patients in this group will have landmark guided arterial line placement.
  Interventions: Procedure: Arterial Line Placement

INTERVENTIONS:
Procedure: Arterial Line Placement — arterial line placement

SUMMARY:
Critically ill patients in the emergency department commonly require arterial line placement for continuous direct blood pressure monitoring, frequent arterial blood gas sampling, and frequent blood sampling. Trans-radial catheterization has been shown to reduce access site complications and increase patient comfort compared to trans-femoral access. Radial artery access on the first attempt is optimal; attempts at reentry delay care and increase the risk of vascular spasm, hematoma, infection, neurovascular injury, and pain. The traditional pulse palpation method of radial artery cannulation can be challenging, especially in patients with weak pulses (i.e. morbidly obese or hypotensive individuals).

A review of literature suggests that ultrasound guided trans-radial catheterization compared to standard pulse palpation reduces access time and increases rate of first-entry success when performed by physicians trained in ultrasound. Thus, complications ascribed to reentry are prevented and timely care is provided.

To the investigator's knowledge, only one other prospective study has been conducted to assess the utility of ultrasound guided radial artery cannulation in the emergency department. Due to the paucity of literature to support the use of ultrasound guided trans-radial catheterization in critically ill patients, the study will aim to provide further data on the topic. Both techniques are considered standard of care.

DETAILED DESCRIPTION:
Patients presenting to the Emergency Department 18 years old or greater, who do not belong to a vulnerable group, requiring arterial line placement will be included in this trial. The investigators will randomize each patient into LM vs US. Data collected will include number of attempts, success rate, and time for procedure to be completed. PGY-1 residents will perform the arterial line placement.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring arterial line placement.

Exclusion Criteria:

* Adults Unable to Consent
* Members of Vulnerable Populations

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Superiority of Method of arterial line placement | 1 day
  Number of attempts until successful cannulation.

SECONDARY OUTCOMES:
Success of method | 1 day
  Completion of arterial line placement after three attempts

CONTACTS AND LOCATIONS:
Overall Officials: Ryan C Gibbons, MD, Principal Investigator — Lewis Katz School of Medicine at Temple University
Locations (1):
- Lewis Katz School of Medicine at Temple University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided